CLINICAL TRIAL: NCT03566043
Title: A Phase 1/2/3 Multicenter, Open-Label Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacodynamics of RGX-121 in Pediatric Subjects With MPS II (Hunter Syndrome)
Brief Title: CAMPSIITE™ RGX-121 Gene Therapy in Subjects With MPS II (Hunter Syndrome)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGX-121-101
Record Dates: First submitted 2018-05-01; First posted 2018-06-21 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Mucopolysaccharidosis Type II (MPS II)
Keywords: MPS II; gene therapy; Hunter Syndrome; Lysosomal Storage Disorder
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death; Lysosomal Storage Diseases

STUDY DESIGN:
Intervention Model Description: Dose escalation
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: RGX-121 Dose 1 (Experimental): 1.3x10^10 GC/g brain mass of RGX-121
  Interventions: Genetic: RGX-121
- Part 1: RGX-121 Dose 2 (Experimental): 6.5x10^10 GC/g brain mass of RGX-121
  Interventions: Genetic: RGX-121
- Part 1: RGX-121 Dose 2 Expanded Cohort (Experimental): 6.5x10^10 GC/g brain mass of RGX-121
  Interventions: Genetic: RGX-121
- Part 1: RGX-121 Dose 3 (Experimental): 2.0x10^11 GC/g brain mass of RGX-121
  Interventions: Genetic: RGX-121
- Part 1: RGX-121 Dose 3 Expanded Cohort (Experimental): 2.9x10^11 GC/g brain mass of RGX-121 (transgene-specific PCR assay) equivalent to, 2.0x10^11 GC/g brain mass of RGX-121 (Poly-A-specific PCR assay)
  Interventions: Genetic: RGX-121
- Part 2: RGX-121 Pivotal Expansion (Experimental): 2.9x10^11 GC/g brain mass of RGX-121 (transgene-specific PCR assay)
  Interventions: Genetic: RGX-121

INTERVENTIONS:
Genetic: RGX-121 — Recombinant adeno-associated virus serotype 9 capsid containing human iduronate-2-sulfatase expression cassette

SUMMARY:
RGX-121 is a gene therapy which is intended to deliver a functional copy of the iduronate-2-sulfatase gene (IDS) to the central nervous system. This study is a safety and efficacy, dose ranging study to determine whether RGX-121 is safe, effective and well-tolerated by patients with MPS II.

DETAILED DESCRIPTION:
MPS II (Hunter Syndrome) is a rare X-linked recessive genetic disease caused by mutations in the iduronate-2-sulfatase gene (IDS). Enzyme replacement therapy (ERT) with recombinant idursulfase (ELAPRASE®) is the only approved product for the treatment of Hunter syndrome, however, ERT as currently administered does not cross the blood brain barrier and is therefore unable to address the unmet need in MPS II patients with central nervous system (CNS) (neurocognition and behavior) involvement. RGX-121 is designed to deliver a functional gene to cells in the CNS. Iduronate-2-sulfatase (I2S) may then be secreted by transduced cells, which may then cross-correct non-transduced cells by taking up the functional enzyme.

This is a Phase I/II/III study enrolling in two sequential parts. Part 1 is a Phase I/II, first-in-human, multicenter, open-label, single arm dose escalation study of RGX-121. Three one-time doses of RGX-121 will be studied in up to 16 pediatric subjects who have neuronopathic MPS II. Safety will be the primary focus for the initial 24 weeks after treatment (primary study period) whereupon, subjects will continue to be assessed (safety and efficacy) for up to a total of 104 weeks following treatment with RGX-121. Part 2 is a pivotal expansion, multicenter, open-label, single arm study of RGX-121. A single dose of RGX-121 will be studied in up to 30 pediatric patients who have been diagnosed with neuronopathic MPS II. Subjects will be assessed at various timepoints for 24 months after receiving RGX-121. Subjects will be given the opportunity to enroll in a separate 3-year long-term follow-up study in accordance with the US federal government guidelines for the safety follow-up of patients receiving gene therapy.

ELIGIBILITY:
Part 1 Inclusion Criteria:

* The subject's legal guardian(s) is (are) willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures
* Is a male ≥4 months to < 5 years of age on Day 1
* Must meet any of the following criteria:

  * Has a documented diagnosis of MPS II and a has a neurocognitive testing score ≤ 77 (Bayley or Kaufman), OR
  * Has a documented diagnosis of MPS II AND has a decline of ≥ 1 standard deviation on serial neurocognitive testing administered between 3 to 36 months apart (Bayley or Kaufman) OR
  * Has a relative clinically diagnosed with severe MPS II who has the same IDS mutation as the subject AND in the opinion of a geneticist has inherited a severe form of MPS II OR
  * Has documented mutation (s) in IDS that in the opinion of a geneticist is always known to result in a neuronopathic phenotype AND in the opinion of a clinician has a severe form of MPS II

Part 2 Inclusion Criteria:

* The subject's legal guardian(s) is (are) willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures
* Is a male ≥4 months to < 5 years of age on Day 1
* Has a documented diagnosis of neuronopathic MPS II. Neuronopathic MPS II can be documented with any of the following methods:

  * Has a BSID-III Cognitive Composite score at or below -1 SD (85) from normative mean
  * Has two consecutive neurodevelopmental assessments that support a decline on MSEL visual receptive, expressive language, or fine motor, or BSID-III cognition, expressive language, or fine motor ≥ 1 SD on serial neurocognitive testing administered between 3 to 36 months apart
  * Has a relative clinically diagnosed with neuronopathic MPS II who has the same IDS mutation as the subject AND the subject, in the opinion of a geneticist, has inherited a neuronopathic form of MPS II
  * Has documented mutation(s) in IDS known to result in a neuronopathic phenotype

Part 1 Exclusion Criteria:

* Has contraindications for intracisternal (IC) injection, intracerebroventricular (ICV) injection or lumbar puncture
* Has contraindications for immunosuppressive therapy
* Has neurocognitive deficit not attributable to MPS II or diagnosis of a neuropsychiatric condition
* Has a (cerebral) ventricular shunt that may impact the proper dosing of the subject
* Received hematopoietic stem cell transplantation
* Has had prior treatment with an AAV-based gene therapy product
* Received ELAPRASE® via intrathecal (IT) administration within 4 months of signing the ICF or experienced a serious hypersensitivity reaction to ELAPRASE®
* Has received any investigational product within 30 days of Day 1 or 5 half-lives before signing the ICF, whichever is longer

Part 2 Exclusion Criteria:

* Has a contraindication for an IC injection, ICV injection or lumbar puncture
* Has contraindications for immunosuppressive therapy
* Has neurocognitive deficit not attributable to MPS II or diagnosis of a neuropsychiatric condition
* Has a (cerebral) ventricular shunt that may impact the proper dosing of the subject
* Received hematopoietic stem cell transplantation
* Has had prior treatment with an AAV-based gene therapy product
* Is receiving idursulfase (ELAPRASE®) via intrathecal (IT) administration, or a blood brain barrier-crossing enzyme replacement therapy. Subjects receiving IT ELAPRASE® or a blood brain barrier-crossing ERT may enroll if they agree to discontinue these therapies starting at least 3 months prior to dosing with RGX-121, and for the 24 months of follow-up
* Has received any investigational product within 30 days of Day 1 or 5 half-lives before signing the ICF, whichever is longer

Ages: 4 Months to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Genetic-based gender identity
Enrollment: 48 (Estimated)
Dates: Start 2018-09-27 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Part 1 Safety | 24 Weeks
  Number of participants with treatment-related adverse events and serious adverse events as assessed by CTCAE (Version 4.03).
Part 2 Biomarkers | 52 Weeks
  CSF GAG levels (as measured by D2S6)
Part 2 Biomarkers | 104 weeks
  CSF GAG levels (as measured by D2S6)
Part 2 Neurodevelopmental parameters | 52 Weeks
  Neurodevelopmental function as measured by the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III) or Mullen Scales of Early Learning (MSEL). The Bayley Scales of Infant Development, or the BSID-III is an individually administered test, designed to evaluate the developmental functioning of infants and small children, between 1 and 42 months of age. The purpose of the test is to identify infants and children with developmental delay. The Mullen Scales of Early Learning (MSEL) is a developmental test to measure cognitive ability, language and motor development. The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. An increase in raw and age equivalent scores indicates neurodevelopmental skill acquisition. Standard scores compare function to age matched normative data.
Part 2 Neurodevelopmental parameters | 104 weeks
  Neurodevelopmental function as measured by the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III) or Mullen Scales of Early Learning (MSEL). The Bayley Scales of Infant Development, or the BSID-III is an individually administered test, designed to evaluate the developmental functioning of infants and small children, between 1 and 42 months of age. The purpose of the test is to identify infants and children with developmental delay. The Mullen Scales of Early Learning (MSEL) is a developmental test to measure cognitive ability language and motor development. The test has five scales: gross motor, visual reception, fine motor, receptive language, and expressive language. An increase in raw and age equivalent scores indicates neurodevelopmental skill acquisition. Standard scores compare function to age matched normative data.

SECONDARY OUTCOMES:
Part 1 Safety | 104 Weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE (Version 4.03)
Part 1 Biomarkers | 104 Weeks
  Glycosaminoglycan levels and iduronate-2-sulfatase activity
Part 1 Neurodevelopmental parameters | 104 Weeks
  Neurodevelopment parameters of cognitive, behavioral & adaptive function as measured by the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III) or Kaufman Assessment Battery for Children, 2nd Edition (KABC-II) and Mullen Scales of Early Learning (MSEL). The BSID-III evaluates the developmental functioning of infants & small children 1 to 42 months old to identify developmental delays. The KABC-II measures cognitive skill & academic knowledge to evaluate knowledge acquired & level of school learning attained. This test evaluates children 2.5 to 12.5 years old in 4 dimensions: mental, sequential and simultaneous processing, & knowledge. The MSEL measures cognitive ability language & motor development & has 5 scales: gross & fine motor, visual reception, & receptive and expressive language. An increase in raw & age equivalent scores indicates neurodevelopmental skill acquisition. Standard scores compare function to age matched normative data.
Part 1 Change in neurodevelopmental parameters | 104 Weeks
  Neurodevelopment parameters of cognitive, behavioral and adaptive function as measured by the Vineland Adaptive Behavior Scales, 2nd Edition (VABS-II), Comprehensive Interview Form. The Vineland Adaptive Behavior Scale II (VABS-II) is a standardized paediatric functional assessment tool. The VABS-II offers a way to measure personal and social self-sufficiency in real-life situations and to observe how these cognitive abilities impact the autonomy management process when put into practice. The VABS-II consists in a semi-structured interview with the parents. Higher scores mean a better outcome.
Part 2 Change in neurodevelopmental parameters | 52 Weeks
  Change from baseline in neurodevelopment effect on daily living skills as measured by the Vineland Adaptive Behavior Scales, 2nd Edition (VABS-II), Comprehensive Interview Form. The Vineland Adaptive Behavior Scale II (VABS-II) is a standardized paediatric functional assessment tool. The VABS-II offers a way to measure personal and social self-sufficiency in real-life situations and to observe how these cognitive abilities impact the autonomy management process when put into practice. The VABS-II consists in a semi-structured interview with the parents. Higher scores mean a better outcome.
Part 2 Change in brain magnetic resonance imaging (MRI) parameters | 52 Weeks
  Change from baseline in brain size as measured on MRI
Part 2 Safety | 24 Months
  Number of participants with treatment-related adverse events as assessed by CTCAE (Version 4.03)
Part 2 Biomarkers | 24 Months
  Change in Glycosaminoglycan levels and iduronate-2-sulfatase activity

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - University of California San Francisco, Benioff Children's Hospital, Oakland, California
  - St. Peter's University Hospital, New Brunswick, New Jersey
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh - UPMC: Program for Neurodevelopment in Rare Disorders, Pittsburgh, Pennsylvania
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No